Analyzing Engagement Trends in Rhabdomyosarcoma Clinical Trials: A Study of Participation Patterns Among Those Affected by the Disorder

An Informed Consent For Patients With Rhabdomyosarcoma in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: September 1, 2023

Information on This Informed Consent Document

If you are tasked with completing this document, it indicates the possibility of your involvement in an observational clinical trial specifically tailored for individuals dealing with rhabdomyosarcoma. This document serves as a comprehensive guide, revealing the study's overarching objectives, intricate execution plan, and multifaceted implications, both positive and potentially otherwise. Delving into the details of your potential participation before making a decision is of utmost importance, and seeking guidance from a trusted source can provide valuable perspectives. Should any aspects of the information contained within this document seem unclear or if questions arise, rest assured that the researcher is readily available to provide clarifications.

Purpose of the Study

Rhabdomyosarcoma is a form of sarcoma. Sarcoma is a kind of cancer that affects soft tissue (like muscle), connective tissue (like tendon or cartilage), or bone. Rhabdomyosarcoma typically starts in muscles that are linked to bones and help the body move, although it can start elsewhere in the body.

Clinical trials tailored to address rhabdomyosarcoma play a pivotal role in assessing the safety and effectiveness of innovative treatments for this condition. These trials are essential in determining whether emerging treatments outperform existing options and provide substantial evidence to support their broader adoption.

This study places a specific focus on delving into the experiences of individuals diagnosed with rhabdomyosarcoma as they actively participate in a unique clinical trial incorporating medical interventions. The primary emphasis centers on closely analyzing trial completion rates and instances of voluntary withdrawal among these participants.

## Exploring the Core of Observational Studies

Participating in this medical trial introduces you to an observational study, a unique aspect of clinical research carefully crafted to glean insights through the unaltered observation of individuals while preserving their care plans.

Researchers will solely focus on observing your journey, meticulously evaluating the outcomes of your condition without making any modifications. This specific trial design plays a pivotal role in enriching our understanding of the inherent progression of a particular medical condition and its effects on those who bear its diagnosis. By actively engaging in this observational study, you contribute significantly to expanding the horizons of medical knowledge and fostering enhancements in the care extended to individuals grappling with the same affliction.

# Distinguishing This Trial from Other Rhabdomyosarcoma Clinical Studies

Recognizing the unique nature of this clinical trial is crucial. It operates within an observational framework, indicating that your involvement won't entail specific treatments or interventions. However, comprehending the full spectrum of rhabdomyosarcoma clinical trials is essential, encompassing interventional studies where participants undergo specific treatment protocols.

Arriving at an informed decision about your possible involvement in a clinical trial necessitates an active approach that includes research and comparison of various studies. Abundant information regarding <u>studies related to rhabdomyosarcoma</u> is accessible through platforms like clinicaltrials.gov. Power's dedicated online platform can give you a comprehensive compilation of ongoing <u>rhabdomyosarcoma clinical trials</u> actively seeking participants. By conducting thorough research and gaining an in-depth

understanding of various clinical trial formats, you empower yourself to form a decision whether you will participate or not.

## Active Participation of Participants

Within the framework of this observational clinical trial, we extend an invitation for you to actively share your experiences. This endeavor involves completion of questionnaires given to you twice a month, necessitating approximately 20-30 minutes of your valuable time. Moreover, at quarterly intervals, we are fully prepared to organize check-in calls, a practice that continues as long as your engagement in the trial persists.

Highlighting its utmost significance, it is essential to underline that your involvement in the survey phase of the trial is entirely voluntary. You can decide whether to address specific questions or the full questionnaire. Furthermore, you maintain the independence to conclude your participation in the trial whenever you see fit. Understanding that the decision to participate in the study is personal, our unwavering commitment is to provide the necessary support. We prioritize your privacy and comfort and we are committed to respecting and supporting your decision-making process throughout the process.

#### Potential Health Concerns

Despite the remarkable progress catalyzed by clinical trials, it's essential to recognize the potential health risks that participants might face, particularly in trials exploring novel treatments.

However, our observational clinical trial follows a different path, proactively addressing these risks by refraining from introducing new interventions to participants. Instead, our primary emphasis lies in thorough observation and measuring outcomes, ensuring that unnecessary health hazards are kept at bay.

#### Potential Positive Outcomes

Although immediate benefits might not be readily apparent for individuals engaging in this observational clinical trial, their participation holds the potential to create a ripple effect. The wealth of data gathered from participants will contribute to refining future methodologies for enrolling rhabdomyosarcoma patients, potentially unlocking broader avenues for medical research. By embarking on this clinical journey, individuals can act as agents of transformative change within the sphere of medical research, potentially redirecting the trajectory for future rhabdomyosarcoma patients.

# Maintaining the Confidentiality of Your Responses

Upholding the utmost confidentiality of your information is of the highest priority during the entire duration of this clinical trial. To protect your anonymity, we respectfully request that you abstain from including any personal or identifiable particulars in your questionnaire responses. The dedicated research team is fully committed to reinforcing the shield of your confidentiality. However, it's important to acknowledge that specific legal circumstances might emerge, necessitating the disclosure of your data.

## Journeying Through Clinical Trial Inclusivity

For those who possess a profound curiosity about exploring the intricate domain of representation in clinical trials, a treasure trove of online resources eagerly awaits your active engagement.

Whether your aspiration is to untangle the complexities of challenges and possibilities surrounding clinical trial diversity or to elevate your personal insights, these sources can serve as enlightening guides:

Le Gal, Frédéric, Ségolène Brichler, Tudor Drugan, Chakib Alloui, Dominique Roulot, Jean-Michel Pawlotsky, Paul Dény, and Emmanuel Gordien. "Genetic diversity and worldwide distribution of the deltavirus genus: a study of 2,152 clinical strains."

Hepatology 66, no. 6 (2017): 1826-1841.

Gomez, Luis Emilio, and Patrick Bernet. "Diversity improves performance and outcomes." *Journal of the National Medical Association* 111, no. 4 (2019): 383-392.

# Confirmation of Voluntary Consent

I affirm that I have devoted substantial time to understand and internalize the content within the informed consent form, either through independent exploration or with the

assistance of a a researcher who explained it to me. All my queries and uncertainties have been answered to my full satisfaction.

I am aware that my participation in this study is the result of my personal decision, and I have the exclusive right to withdraw my permission at any time.

Having diligently contemplated and evaluated the form presented to me, I hereby provide my agreement to join this clinical trial, reflecting my well-informed and self-governing choice.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| Date |

# Confirmation by Informed Consent Facilitator

I hereby confirm that I have engaged in a dialogue with the participant, explaining the entirety of this written document. My primary goal was to ensure that the participant comprehended the trial's objectives, processes, potential risks and benefits, as well as other factors intrinsic to the clinical trial centered around rhabdomyosarcoma.

The participant was given adequate inquiry space, which encouraged the formation of questions and facilitated the explanation of ambiguities or misconceptions. It is critical to underline that the participants' participation in this trial is the result of their voluntary decision, and they have the ultimate right to withdraw at any time, for any reason, without incurring any financial responsibilities.

A duplicate of this written document was supplied to them, serving as a reference for future use.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| <br>Date |